CLINICAL TRIAL: NCT04392063
Title: Effect of Melatonin Supplementation on Sleep and Health of Children With Cerebral Palsy
Brief Title: Melatonin for Cerebral Palsy Children's Sleep and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sahar M.A. Hassanein, MD, Professor of Pediatrics, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 202/2016
Record Dates: First submitted 2020-05-10; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Cerebral Palsy; Melatonin; Growth; Children, Only
Keywords: Children's sleep habits questionnaire (CSHQ) Arabic version; Anthropometry; GERD; Constipation; Polysomnography
MeSH Terms: conditions — Cerebral Palsy; Gastroesophageal Reflux; Constipation | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: A prospective, cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerebral palsy (Other): Not included
  Interventions: Drug: Melatonin 3 mg

INTERVENTIONS:
Drug: Melatonin 3 mg — The children received crushed Melatonin 3-mg tablets daily, 30-minutes before bedtime for 3-months.
  Other Names: Melatonin CP

SUMMARY:
The present study was prospective uncontrolled, single-armed and un-blinded study. Held in the Pediatric neurology clinic, Children's hospital l, Faculty of Medicine, Ain Shams University from June 2016 to June 2018 of 24 months timeframe. All cerebral palsy (CP) patients following up in Pediatric neurology clinic aged between 2 and 12 years. Melatonin given for 3 months. Anthropmetric measures, gastroeintestinal symptoms, Children's sleep habits questionnaire (CSHQ) Arabic version, polysomnography, Chalfont epilepsy severity score, and EEG were done at enrollment and after the 3-months.

DETAILED DESCRIPTION:
A prospective, cohort study conducted in Pediatric Neurology Clinic, Children's Hospital, Faculty of Medicine, Ain Shams University. Forty children with sCP with sleep and seizure problems, aged 2-12 years were enrolled. The children received crushed Melatonin 3-mg tablets daily, 30-minutes before bedtime for 3-months. Children's sleep habits questionnaire (CSHQ) Arabic version, polysomnography, Chalfont epilepsy severity score, and EEG were done at enrollment and after the 3-months. The ethical approval number is (FMASU MD 202/2016).

ELIGIBILITY:
Inclusion Criteria:

* All cerebral palsy children with sleep problem and seizure disorder,
* aged 2 - 12 years

Exclusion Criteria:

* any auditory and peripheral visual impairments

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Decrease in total Children's sleep habits questionnaire score | after 3-months
  response to melatonin as decrease in total sleep score
Improvement in growth | 3-months
  response to melatonin in improvement of growth

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elkhayat HA, Hassanein SM, Tomoum HY, Abd-Elhamid IA, Asaad T, Elwakkad AS. Melatonin and sleep-related problems in children with intractable epilepsy. Pediatr Neurol. 2010 Apr;42(4):249-54. doi: 10.1016/j.pediatrneurol.2009.11.002. PMID 20304327
- See also: Published part of the work "Effect of Melatonin Supplementation on Gastrointestinal Problems and Growth of Children with Cerebral Palsy" — https://platform.almanhal.com/Reader/Article/130441